CLINICAL TRIAL: NCT02480088
Title: Comparison of Palonosetron and Ramosetron for Preventing Patient-controlled Analgesia Related Nausea and Vomiting Following Spine Surgery; Association With ABCB1 Polymorphism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2014-0583
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ramosetron; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ramosetron (Experimental): patients receiving ramosetron for prophylaxis of postoperative nausea and vomiting
  Interventions: Drug: Ramosetron
- palonosetron (Active Comparator): patients receiving palonosetron for prophylaxis of postoperative nausea and vomiting
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Ramosetron — ramosetron 0.3 mg IV 20 min before the end of surgery and 24 h after the surgery
  Arms: ramosetron
Drug: Palonosetron — palonosetron 0.075 mg IV 20 min before the end of surgery and 24 h after the surgery.
  Arms: palonosetron

SUMMARY:
Opioid-based intravenous patient-controlled analgesia (IV-PCA) offers excellent pain control, however, its use inevitably increases the incidence of postoperative nausea and vomiting (PONV). Ramosetron and palonosetron are commonly used 5-HT3 antagonists for the prevention and treatment of PONV. It is not clear which one has superior antiemetic efficacy for the prevention of PONV in patients using opioid-based IV-PCA. The antiemetic efficacy of 5HT3 antagonists may be influenced by polymorphism of ABCB1, a drug-transporter gene. This study evaluates relative antiemetic efficacy of ramosetron and palonosetron in patients using IV-PCA after spinal surgery and impact of ABCB1 polymorphism on the antiemetic efficacy of the ramosetron and palonosetron. The incidence and intensity of PONV during postoperative 48 h will be assessed. ABCB1 polymorphisms 3435C>T and 2677G>T/A will be evaluated in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-85 yr
* undergoing spine surgery

Exclusion Criteria:

* Taking steroids or opioids preoperatively
* GI motility disorder
* Uncontrolled diabetes
* Severe renal or hepatic disease
* Transfer to ICU postoperatively
* Obesity (BMI>35 kg/m2)
* Use of antiemetic agent within 24 h preoperatively
* Pregnancy
* Psychiatric disease
* Drug or alcohol abuser
* Malignancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2015-03-11 (Actual); Study Completion 2015-03-11 (Actual)

PRIMARY OUTCOMES:
number of postoperative nausea and vomiting incidence | during postoperative 48h

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia, Seoul, South Korea